CLINICAL TRIAL: NCT06530108
Title: The Effect of Sexual Education Based on the PLISSIT Model on Sexual Function, Attitudes Towards Sexuality and Sexual Distress in Pregnant Women
Acronym: Pregnant Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Esma Demirezen, assistant professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-74555795-199-990466 17.05.24; 17.05.2024-990466 (Other: ISTANBUL UNIVERSITY)
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Healthy; Pregnancy Related; Stress
Keywords: sexual function; sexual attitude; sexual distress; midwife care; education

STUDY DESIGN:
Intervention Model Description: The research will be conducted using randomized controlled, experimental type and single-blindresearch methods. For this purpose, after the data are collected, they will be coded as A and Bgroups, so the researcher who will make the research statistics will analyze the data withoutknowing the study and control groups. Randomization method will be used to determine thegroups. For this, the patients who meet the study criteria and volunteer will be assigned to thegroups using the randomization program 'Random Allocation Software 2.0' according to the orderof hospitalization.
Who Masked: Participant
Masking Description: The data analyse is going to be completed by a independent researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention Group (Experimental): PLISSIT model-based sexual health education will be provided to the intervention group, and the clinical procedure will be applied to the control group. The Sexual Attitude Scale during Pregnancy and the Female Sexual Distress Scale will be administered simultaneously. Four weeks after the training, the FSFI application and the Sexual Attitude Scale during Pregnancy and the Female Sexual Distress Scale will be administered again
  Interventions: Behavioral: PLISSIT model based sexual health education
- Kontrol Group (Placebo Comparator): The clinical procedure will be applied to the control group
  Interventions: Behavioral: PLISSIT model based sexual health education

INTERVENTIONS:
Behavioral: PLISSIT model based sexual health education — the PLISSIT model includes the steps of PLISSIT (P-Permission), LI-Limited Information, SS-Specific Suggestions, IT-Intensive Therapy. This model provides communication with the patient and Since it is a model that increases confidence and provides care interventions based on the patient's preference, it has the feature of guiding sexual education during pregnancy by establishing the bond between the pregnant woman and the midwife.

SUMMARY:
The Effect of Sexual Education Based on the PLISSIT Model on Sexual Function, Attitudes towards Sexuality and Sexual Distress in Pregnant Women

Purpose of the study: In the light of these data, the effect of sexual health education based on the PLISSIT model on sexual function, attitude towards sexuality and sexual distress in nulliparous pregnant women will be examined in a randomized controlled experimental study. It is thought that the data to be obtained will shed light on sexual health education and counseling practices for midwives working with pregnant women in their application areas.

DETAILED DESCRIPTION:
The Effect of Sexual Education Based on the PLISSIT Model on Sexual Function, Attitudes towards Sexuality and Sexual Distress in Pregnant Women

Method of the study: FSFI will be applied to pregnant women between 14-20 weeks of gestation who apply to Trakya University Health Research and Application Center Obstetrics Clinic, Polyclinic and Perinatology Clinic departments, and women with a score ≤ 26.55 as a result of the FSFI evaluation will be defined as having sexual dysfunction. Pregnant women will be randomized according to the last digit of their protocol number. Pregnant women divided into control and intervention groups will be given PLISSIT model-based sexual health education to the intervention group and a clinical procedure will be applied to the control group. The Sexual Attitude Scale during Pregnancy and the Female Sexual Distress Scale will be administered simultaneously. Four weeks after the training, the FSFI application and the Sexual Attitude Scale during Pregnancy and the Female Sexual Distress Scale will be administered again.

ELIGIBILITY:
inclusion criteria: Volunteer to participate, 19 years of age and over, sexually active, at least primary school graduate, of Turkish origin, no communication problems, 14th-20th age, fluent in Turkish. Pregnant women in their 2nd week will be included in the study.

exclusion criteria: Pregnant women who are at serious risk during pregnancy, who are diagnosed with sexual dysfunction, who have mental problems that require treatment, and who use drugs that cause sexual dysfunction will not be included in the study Pregnant women who leave their information forms unfinished, experience loss, and want to leave the study will be excluded.

-

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant Women
Enrollment: 180 (Estimated)
Dates: Start 2024-05-18 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Sexual Function Level | 12 Mounth
  Women with a score ≤ 26.55 as a result of the FSFI evaluation will be defined as having sexual dysfunction.

SECONDARY OUTCOMES:
Attitude Towards Sexuality During Pregnancy | 12 mounth
  An increase in the Attitude Towards Sexuality During Pregnancy score indicates that attitudes towards sexuality during pregnancy are positive.
Sexual Distres Level | 12 mounth
  KCDÖ-R consists of 13 items that evaluate different aspects of sexual distress in women and varies between 0-52 points. The scale is a five-point Likert type and is scored between 0-4 points (always=4, often=3, sometimes=2, rarely=1, never=0), and 11.5 and above is defined as sexual distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No